CLINICAL TRIAL: NCT04798898
Title: Improving Survival of COlorectal LIver Metastases by RFA-mediated Immunostimulation
Acronym: ISCOLIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISCOLIM
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Liver Metastasis Colon Cancer
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (+RFA) arm (Experimental): Preoperative partial RFA necrosis in the liver metastasis followed by liver resection
  Interventions: Device: RFA (radiofrequency ablation)
- Control (-RFA) arm (No Intervention): Liver resection

INTERVENTIONS:
Device: RFA (radiofrequency ablation) — Preoperative RFA-induced partial necrosis of the liver metastasis
  Arms: Intervention (+RFA) arm

SUMMARY:
To examine radio frequency ablation as a treatment supplement to stimulate immunogenicity and improve survival for patients undergoing curative-intent surgery for colorectal liver metastases.

DETAILED DESCRIPTION:
PURPOSE:

To investigate the impact of immunostimulation using radio frequency ablation (RFA) on survival in patients undergoing curative-intent surgery for colorectal liver metastases (CRLM).

HYPOTHESIS:

RFA-mediated partial destruction of CRLM will stimulate the immune system to recognize otherwise hidden cancer antigens, which in turn will improve survival by inhibiting micrometastases and recurrence.

BACKGROUND:

CRLM affects around 1,600 individuals in Denmark each year. State-of-the-art treatment includes liver resection, RFA treatment, radiation therapy, and chemotherapy. Of all individuals undergoing surgery, 50% will experience local or distant recurrence of the disease within five years. Although liver resection is the gold standard, RFA treatment has evolved considerably in recent years. RFA is a parenchymal-sparing treatment for hepatic malignancies, inducing a localized coagulation necrosis of the tumor. This leads to release of tumor antigens, which activates the patients' immune system. However, many cancer cells, including those from CRLM, have the ability to hide their antigens to the patients' immune systems. Using RFA as immunostimulation prior to surgery, these antigens may become visible to the immune system, which in turn can help eradicating all tumor cells and decrease the risk of tumor recurrence. Combined, this likely improves survival.

METHODS:

220 patients with CRLM planned for surgery will be enrolled in this study. Patients will be randomized to +/- RFA treatment before surgery. Under guidance of ultrasonography, a single-electrode RFA-needle is placed in a CRLM with a diameter of at least 3 cm, which is later going to be resected. In 20 of the patients, we will draw blood samples for determination of immune status both pre- and postoperatively. All patients will be part of a work-up with regular CT-scans.

ENDPOINTS:

Disease free survival and overall survival. Secondarily, we will examine the effect of RFA treatment of tumors on the innate and adaptive immune system in 20 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal liver metastases planned for resection
* At least one tumor size >=3cm
* Performance status 0-1

Exclusion Criteria:

* Liver cirrhosis
* Extrahepatic metastases that can not be addressed curatively
* Other malignant diseases within 5 years prior to diagnosis
* Prior RFA treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  Median survival in each arm

SECONDARY OUTCOMES:
One-year survival | 1 year
  One-year survival in each arm
Two-year survival | 2 years
  Two-year survival in each arm
Three-year survival | 3 years
  Three-year survival in each arm
Recurrence rate | 1, 2, and 3 years
  Recurrence rate at 1, 2, and 3 years follow-up

OTHER OUTCOMES:
Complications | 30-day postoperatively
  Immediate postoperative complications (bleeding, surgical site infection, intraabdominal abscesses, bile leak)

CONTACTS AND LOCATIONS:
Overall Officials: Frank V Mortensen, MD, DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Surgery, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04798898/Prot_SAP_001.pdf